CLINICAL TRIAL: NCT05712343
Title: The Efficacy of Systemic Valacyclovir (Valtrex) to Arrest Further Progression of Severe Periodontitis
Brief Title: The Efficacy of Systemic Valacyclovir (Valtrex) on Periodontitis
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 22-36008
Record Dates: First submitted 2023-01-25; First posted 2023-02-03 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Severe Periodontitis
MeSH Terms: conditions — Periodontitis | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- valacyclovir group (Experimental): Patients (N=20) in the valacyclovir group will be received, at baseline, periodontal scaling + valacyclovir (500 mg, 3 times a day for 3 days) ("Valacyclovir" group).
  Interventions: Drug: Valacyclovir group
- Control group (Active Comparator): Patients (N=20) in the control group will receive, at baseline, periodontal scaling + placebo medication, three times a day for 3 days ("Control" group).
  Interventions: Other: Control group

INTERVENTIONS:
Drug: Valacyclovir group — The valacyclovir group will be received, valacyclovir (500 mg, 3 times a day for 3 days)
  Arms: valacyclovir group
Other: Control group — The control group will receive placebo medication, three times a day for 3 days.
  Arms: Control group

SUMMARY:
The experiment outlined in this proposal is designed to test the hypothesis that herpesvirus suppression by the systemic anti-herpesvirus valacyclovir (Valtrex) can significantly help to arrest the progressive course of severe marginal periodontitis in adult patients. A prospective, randomized, placebo-controlled, double-blind, clinical trial is employed to test this hypothesis.

DETAILED DESCRIPTION:
This study will be conducted as a double-blind, randomized, 6-month clinical trial to test the efficacy of systemic valacyclovir to prevent further progression of severe periodontitis. Subjects with at least 4 deep vertical periodontal lesions (> 4 mm loss of clinical attachment level) showing no radiographic crestal alveolar lamina dura will be randomly assigned to one of two treatment groups. Patients (N=20) in the valacyclovir group will be received, at baseline, periodontal scaling + valacyclovir (500 mg, 3 times a day for 3 days) ("Valacyclovir" group).

Patients (N=20) in the control group will be received, at baseline, periodontal scaling + placebo medication, three times a day for 3 days ("Control" group). All patients in both treatment groups will be evaluated for the status of their periodontal disease after 3 months by assessing clinical attachment level changes, periodontal pocket depth, and gingival bleeding on probing. Patients showing one or more periodontal site(s) with ongoing clinical attachment level loss of 2 mm or more will be exited from the study and receive conventional periodontal treatment such as systemic antibiotics or surgery. Patients demonstrating no additional clinical attachment level loss will remain in the study for another 3 months, after which a final assessment of the periodontal status will be performed as described above. All patients will then be referred for conventional periodontal treatment. Using a random number generator, patients will be assigned to a study group and given an undifferentiable, opaque Manila packet containing valacyclovir or placebo medication as well as written instructions. Oral hygiene instructions will be given to all subjects at baseline by a dental hygienist. Follow-up oral hygiene evaluation and instruction and dental plaque recording will be performed at 3- and 6-months post baseline treatment by a dental hygienist. Study patients will be provided with one 8 oz toothpaste (Regular Colgate) and a soft toothbrush (Oral-B Soft). Patients will need to sign informed consent before enrollment into the study. Patients are free to discontinue the study at any time for any or for no reason. A periodontist who is blinded to the baseline valacyclovir/placebo treatment will perform the clinical and radiographic diagnostic procedures. Clinical examinations, carried out at baseline and at 3-and 6-month post-baseline treatment, will include a whole-mouth measurement of clinical attachment loss level, periodontal pocket depth, plaque index and degree of gingivitis (bleeding on probing). Radiographic evaluation of alveolar bone level and appearance (presence or absence of radiographic crestal alveolar lamina dura) will be performed at baseline and at 6- month post-treatment. The Mann-Whitney statistical tests will assess the outcome data. A manageable patient sample size of 40 is estimated to detect, with a power of 80% and a type I error of 0.05, a difference in periodontal outcome between the valacyclovir and the placebo group. A statistician will analyze the data.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be systemically healthy, Class I dental category.
* Involved teeth must have periodontal disease detectible by periodontal examination.
* Subjects with deep vertical periodontal lesions (>6 mm) showing no radiographic crestal alveolar lamina dura

Exclusion Criteria:

* Presence of any disease or medication that alters the immune system or interferes with healing ability Smokers (more than 10 cigarettes per day)
* External or internal tooth resorption
* Tooth perforation from the pulp cavity through the tip of the root exposing the tissue to material in the oral cavity.
* Pregnant or nursing mothers because hormonal factors may influence the condition.
* Allergies or adverse reactions to valacyclovir.
* Patients under the age of 18.
* Patients with renal impairment or reduced renal function.
* Patients requiring hemodialysis or peritoneal dialysis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-05-25 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Clinical attachment level | 6 months
  Clinical examinations, carried out at baseline and at 3-and 6-month post-baseline treatment, will include a whole-mouth measurement of clinical attachment loss level
Periodontal pocket depth | 6 months
  Clinical examinations, carried out at baseline and at 3-and 6-month post-baseline treatment, will include a whole-mouth measurement of periodontal probing depth
gingival bleeding on probing | 6 months
  Clinical examinations, carried out at baseline and at 3-and 6-month post-baseline treatment, will include a whole-mouth measurement of gingival bleeding on probing

CONTACTS AND LOCATIONS:
Overall Officials: Mike Sabeti, DDS, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Herpesviral-bacterial interactions in periodontal diseases — https://pubmed.ncbi.nlm.nih.gov/20017799/
- See also: Herpesviruses in periodontal diseases — https://pubmed.ncbi.nlm.nih.gov/15853936/